CLINICAL TRIAL: NCT04051151
Title: Move to Improve Physical Activity in Parkinson's Disease: MoTIvatE PD
Brief Title: Move to Improve Physical Activity in Parkinson's Disease
Acronym: MoTIvatE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Nabila Dahodwala, MD, Associate Professor of Neurology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MoTIvatEPD
Record Dates: First submitted 2019-07-26; First posted 2019-08-09 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Parkinson Disease; Apathy
Keywords: Physical Activity; Social Incentives; Behavioral Economics; Goal-Directed Behavior; Motivation
MeSH Terms: conditions — Parkinson Disease; Lethargy; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gameification Arm (Experimental): Participants and partners that have randomized to the gamification group will receive instructions and help in setting up a game.
  Interventions: Behavioral: Gameficiation
- Education Arm (No Intervention): Participants and partners that randomized to the control group will receive standard of care educational resources on the importance of physical activity in Parkinson's patients.

INTERVENTIONS:
Behavioral: Gameficiation — Participants and partners that have randomized to the gamification group will receive instructions and help in setting up a game platform via Way to Health. This game will include wearing a Fit Bit device, setting a daily step goal, and point deductions for failure to meet this step goal throughout the following 4 weeks. Participants will move up or down specified levels each week depending on how many days they met their step goal.
  Arms: Gameification Arm

SUMMARY:
Apathy is a multi-dimensional behavior characterized by impairments to motivation, planning and initiation; collectively called, goal-directed behavior. It is highly prevalent in patients suffering from neurological disorders such as Alzheimer's disease and Parkinson's disease (PD) as well as psychiatric disorders such as depression and schizophrenia. In PD, specifically, apathy is one of the more troublesome symptoms. Apathetic PD patients have greater disability, lower adherence to treatment plans and caregivers report greater stress and burden.

Interventions grounded in behavioral economic theories, namely, financial and social incentives often promote positive behavioral change such as weight loss and smoking cessation. However, the effectiveness of these interventions varies across and within conditions and incentive type. It also tends to dissipate when incentives are no longer provided. To date, these approaches have not been used to promote behavior change in PD or other neurological conditions where apathetic behaviors are a pressing problem. The overall goal of this study is to test if behavioral economic approaches will reduce apathy, and subsequently, improve goal-directed behavior in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will have a diagnosis of Parkinson's disease, and may have either normal cognition or mild cognitive impairment (MCI). Most eligible participants will have to have smartphones with wifi, application, Bluetooth, and text messaging capabilities. The study team does have five smart phone that can be provided to participants who do not have smartphones so as to not exclude these individuals.
* Eligible participants will have to be mobile as the primary outcome measure for the study is step goals measured on the Fitbit. Participants will be eligible if they can ambulate successfully with a cane.
* Participants will also need a study partner to be eligible to participant. This partner can be anyone of the eligible participant's choosing, who also consents to participation in the study.

Exclusion Criteria:

* Individuals will be excluded if they screen positive for dementia at the screening visit or do not have the decisional capacity to give consent. Dementia will be defined as a Montreal Cognitive Assessment (MoCA) score of <22. Decisional capacity will be tested based on their understanding of study risks and benefits.
* Individuals will also be excluded if they require a wheelchair or walker, or are unable to ambulate safely.
* Individuals will be excluded if they are currently participating in another physical activity study, have been told by a physician not to exercise, or are currently pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of gameification intervention to improve physical activity levels | Four weeks
  To test the feasibility and preliminary effectiveness of a gamification intervention that enhances supportive social incentives that includes collaboration, accountability and peer support to improve physical activity levels compared to a control group that receives the standard of care. The researchers will compare the change in mean daily steps between the gameification and control (education) groups using an independent t-test.
Ability of behavioral phenotyping to predict step goal achievement | Four weeks
  Among participants in the intervention group, the researchers will compare the number of days that step goals were achieved between individuals with greater motivation deficits and those with initiation and planning deficits using a one-way independent ANOVA.
Ability of behavioral phenotyping to predict change in activity | Four weeks
  Among participants in the intervention group, the researchers will compare the change in mean daily steps between individuals with greater motivation deficits and those with initiation and planning deficits using a one-way independent ANOVA.

CONTACTS AND LOCATIONS:
Overall Officials: Nabila Dahodwala, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania's Parkinson's Disease and Movement Disorder Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy R, Dubois B. Apathy and the functional anatomy of the prefrontal cortex-basal ganglia circuits. Cereb Cortex. 2006 Jul;16(7):916-28. doi: 10.1093/cercor/bhj043. Epub 2005 Oct 5. PMID 16207933
- [Background] Starkstein SE, Mayberg HS, Preziosi TJ, Andrezejewski P, Leiguarda R, Robinson RG. Reliability, validity, and clinical correlates of apathy in Parkinson's disease. J Neuropsychiatry Clin Neurosci. 1992 Spring;4(2):134-9. doi: 10.1176/jnp.4.2.134. PMID 1627973
- [Background] Pedersen KF, Larsen JP, Alves G, Aarsland D. Prevalence and clinical correlates of apathy in Parkinson's disease: a community-based study. Parkinsonism Relat Disord. 2009 May;15(4):295-9. doi: 10.1016/j.parkreldis.2008.07.006. Epub 2008 Sep 17. PMID 18801696
- [Background] Leiknes I, Tysnes OB, Aarsland D, Larsen JP. Caregiver distress associated with neuropsychiatric problems in patients with early Parkinson's disease: the Norwegian ParkWest study. Acta Neurol Scand. 2010 Dec;122(6):418-24. doi: 10.1111/j.1600-0404.2010.01332.x. PMID 20175757